CLINICAL TRIAL: NCT00166426
Title: Prospective, Randomized, Double-Blind Trial of Adjuvant Exisulind Versus Placebo for Patients at Risk for Prostate Cancer Recurrence After Radical Prostatectomy
Brief Title: Exisulind Versus Placebo After Surgical Removal of the Prostate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: OSI Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 526-02
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2009-11-16 (Estimated); Status verified 2009-11

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sulindac sulfone

INTERVENTIONS:
Drug: Exisulind

SUMMARY:
This is a study in which patients with prostate cancer treated by surgical removal of the prostate and considered to be at risk for prostate cancer recurrence will receive Exisulind 250 mg twice a day or placebo twice a day for two years.

ELIGIBILITY:
Males 18 years of age or older with prostate cancer treated primarily by radical prostatectomy and randomized within 45 days after surgery may be eligible for enrollment into this protocol. Participants cannot have had hormonal therapy, cryotherapy, thermotherapy, or radiotherapy prior to entering the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2003-02; Primary Completion 2007-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Assess efficacy of drug vs placebo regarding overall rate of biochemical progression
Assess the efficacy of drug vs placebo regarding time to biochemical progression
Assess efficacy of drug vs placebo regarding overall rate of clinical progression
Assess efficacy of drug vs placebo regarding time to clinical progression
Assess efficacy of drug vs placebo regarding cancer specific survival

CONTACTS AND LOCATIONS:
Overall Officials: Bradley C. Leibovich, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States